CLINICAL TRIAL: NCT01323400
Title: A Phase II Randomized Multicentre Study Evaluating the Efficacy of Pazopanib+Best Supportive Care (BSC) Versus BSC Alone in Metastatic and/or Locally Advanced Unresectable GIST, Resistant to Imatinib and Sunitinib
Brief Title: Efficacy of Pazopanib in Gastrointestinal Stromal Tumors (GIST)
Acronym: PAZOGIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAZOGIST
Record Dates: First submitted 2011-03-10; First posted 2011-03-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: GIST
Keywords: GIST; Resistant; Pazopanib; Tyrosine kinase inhibitor; Best supportive care; Progression-free survival; Overall survival; Objective response rate; Best response; Tolerance profile
MeSH Terms: interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pazopanib (Experimental): Pazopanib (800 mg/day) + Best supportive care according to the investigator's judgement.
  Pazopanib treatment is started on the day after randomization until radiological progression according to RECIST or until documented toxicity. In case of radiological progression, pazopanib may be continued (if the investigator wishes so) if a clinical benefit (pain reduction, 1 point increase in performance status) is observed.
  Interventions: Drug: Pazopanib; Other: Best supportive care
- Best supportive care (Other): Best supportive care according to the investigator's judgment. Upon progression, compassionate treatment by pazopanib is possible according to eligibility criteria.
  Interventions: Other: Best supportive care

INTERVENTIONS:
Drug: Pazopanib — Pazopanib is administered orally at 800 mg/day (one dose every morning). A dose modification is possible in case of documented toxicity, according to specific algorithms.
  Arms: Pazopanib
Other: Best supportive care — Best supportive care according to the investigator's judgment (chemotherapy, immunotherapy, hormone therapy are not allowed).
  Non-targeted radiation therapy is tolerated, as antalgic strategy. Surgery is tolerated in case of emergency.

SUMMARY:
The purpose of this study is to evaluate the antitumor activity of pazopanib in patients with metastatic and/or locally advanced unresectable Gastrointestinal Stromal Tumors (GIST) resistant to imatinib and sunitinib. This is a phase II, randomized, multicentre study.

DETAILED DESCRIPTION:
Complete resection, with or without associated anticancer therapy, is the standard treatment of GIST. Even though the prognosis of advanced GIST has been tremendously improved by the introduction of tyrosine kinase inhibitors (TKI-imatinib, sunitinib...), the vast majority of patients will develop secondary resistance to these agents. The therapeutic options for patients with advanced GIST with resistance (or intolerance) to imatinib and sunitinib remain very limited. Some new molecules are currently being evaluated in patients with metastatic or locally advanced - imatinib-resistant disease. Nilotinib, for instance, has been evaluated in phase I/II trials and compassionate use programs with a median progression-free survival (PFS) close to 3 months and a median overall survival close to 8.5 months. A phase III trial comparing nilotinib vs. best supportive care (BSC) +/- imatinib or sunitinib (investigators choice) has just been completed and results are pending. Another molecule, Sorafenib, has been evaluated in 4th line treatment in compassionate use studies, with a median PFS close to 5 months and a median overall survival of 10-13 months. There are currently no recognized standard options after failure of 2nd line treatment, and the recently updated guidelines from the NCCN or ESMO (2009) suggest the possible reintroduction of TKI in an attempt to control the progression of sensitive cell clones.

Pazopanib is a broad spectrum TKI targeting KIT, PDGFR and VEGFR which has been tested in phase II trials in advanced sarcomas and has demonstrated promising antitumor activity. Whether pazopanib would be useful in patients with GIST is not known.

In the present study, we propose to analyze the antitumor activity of pazopanib in patients with GIST refractory to imatinib and sunitinib. The drug will be tested against BSC in a randomized setting, with possible crossing-over to the no-treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically confirmed, unresectable, metastatic and/or locally advanced GIST.
3. Progression or intolerance after treatment with at least imatinib (400 mg and 600/800 mg/d) then sunitinib at either 50mg/d on a 4w/6w schedule or 37.5mg/d continuous dosing. Intolerance is defined as documented grade 3 or higher toxicity requiring treatment interruption as documented in patient record.
4. Measurable disease according to RECIST v1.1.
5. Performance status ≤ 2 (WHO).
6. Left Ventricular Ejection Fraction (LVEF) in accordance with local standards.
7. Adequate organ system functions as defined below:

   * Haematologic parameters

     * Absolute neutrophil count (ANC) ≥ 1.5 G/L
     * Haemoglobin ≥ 9 g/dL
     * Platelets ≥ 100 G/L
     * Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.2 X upper limit of normal (ULN) NB: Subjects receiving anticoagulation therapy are eligible if INR is stable and within the recommended range.
     * Partial thromboplastin time (PTT) ≤ 1.2 X ULN
   * Hepatic parameters

     * Total bilirubin ≤ 1.5 X ULN
     * AST and ALT ≤ 2.5 X ULN
   * Renal parameters

     * Serum creatinine ≤ 1.5 mg/dL (133 µmol/L) or, if greater than 1.5 mg/dL: calculated creatinine clearance ≥ 50 mL/min
     * Urine Protein to Creatinine ratio (UPC) < 1. If UPC ≥ 1, subjects must have a 24-hour urine protein value <1g to be eligible.
   * Biochemical parameters

     * Kaliemia ≥ 1 X lower limit of normal (LLN)
8. a) Females of non-childbearing potential (i.e., physiologically incapable of becoming pregnant).

   b) Females of childbearing potential provided that they are not pregnant or lactating, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and who agrees to use adequate contraception.
9. Affiliation with a health insurance company.
10. Subjects must provide written informed consent

Exclusion Criteria:

1. Prior malignant disease (other than GIST) within 3 years prior to entry, with the exception of in situ breast cell carcinoma or in situ carcinoma of the cervix or basocellular carcinoma or spinocellular carcinoma or bladder neoplasm, treated at least 6 months before and with no evidence of relapse.
2. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for patients with previously-treated CNS metastases, who are asymptomatic and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. CNS screening with computed tomography [CT] or magnetic resonance imaging [MRI] is required only if clinically indicated or if the subject has a history of CNS metastases.
3. Treatment with any of the following anti-cancer therapies:

   * radiation therapy, surgery or tumour embolisation within 14 days prior to the first dose of pazopanib OR
   * chemotherapy, biological therapy or investigational therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib.

   The analgesic radiation therapy is allowed (the irradiated lesions won't be chosen as target lesions during the evaluation)
4. Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 followed and/or progressing in severity, except alopecia.
5. Other uncontrolled severe medical conditions.
6. Presence of uncontrolled infection.
7. Clinically significant gastrointestinal abnormalities

   * that may increase the risk for gastrointestinal bleeding.
   * that may affect absorption of investigational product.
8. Poorly controlled hypertension [defined as systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg].

   NB: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions at > 1 hour interval; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <140/90 mmHg for the subject to be eligible to the study.
9. History of any cardiovascular pathology within the past 6 months.
10. Corrected QT interval (QTcB) > 480 msec using Bazett's formula.
11. History of cerebrovascular accident, including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT), within the past 6 months.

    NB: Subjects with recent DVT treated with therapeutic anti-coagulating agents at least 6 weeks before inclusion are eligible.
12. Major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture or ulcer (procedures such as catheter placement are not considered to be major).
13. Evidence of active bleeding or bleeding diathesis.
14. Haemoptysis within 8 weeks before inclusion.
15. Platelet transfusion in the past 7 days.
16. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
17. Concomitant bilirubin and AST/ALT elevations above ULN.
18. Treatment with anti-vitamin K (LMWH are allowed).
19. Inability or unwillingness to discontinue prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
20. Inability to swallow.
21. Pregnant or lactating woman
22. Impossibility to comply with protocol constraints

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Within 16 months after the first inclusion, from the date of randomisation until the date of the first documented progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | Within 16 months after the first inclusion, from the date of randomisation until the date of death from any cause
Objective tumour response rate (RECIST v.1.1) at 4 months | 4 months after randomisation
Best response (RECIST v.1.1) obtained during the study | Within 16 months after the first inclusion
Tolerance profile (NCI-CTCAE v.4.0) | Within 16 months after the first inclusion
Pattern of progression-free survival in the different molecular subtypes | Within 16 months after the first inclusion, from the date of randomisation until the date of the first documented progression or death from any cause
Intra and inter-patient variability of the Cmin of pazopanib | After 4 weeks, 10 weeks, 16 weeks of pazopanib treatment and at time of progression
Progression-free survival in patients not randomly assigned to pazopanib, but receiving pazopanib on a compassionate basis after progression | Within 16 months after the first inclusion, from the date of the first pazopanib administration until the date of the first documented progression or death from any cause
Overall survival in patients not randomly assigned to pazopanib, but receiving pazopanib on a compassionate basis after progression | Within 16 months after the first inclusion, from the date of the first pazopanib administration until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, MD, Principal Investigator — Centre Léon Bérard, LYON, FRANCE
Locations (13):
- France (13):
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Institut Paoli Calmette, Marseille
  - Centre Alexis Vautrin, Nancy
  - Institut de Cancérologie de l'Ouest, Nantes
  - Hôpital St Antoine, Paris
  - Hôpital Tenon, Paris
  - CHU de Reims, Reims
  - Institut Cancerologie Neuwirth, Saint-Priest-en-Jarez
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blay JY, Bonvalot S, Casali P, Choi H, Debiec-Richter M, Dei Tos AP, Emile JF, Gronchi A, Hogendoorn PC, Joensuu H, Le Cesne A, McClure J, Maurel J, Nupponen N, Ray-Coquard I, Reichardt P, Sciot R, Stroobants S, van Glabbeke M, van Oosterom A, Demetri GD; GIST consensus meeting panelists. Consensus meeting for the management of gastrointestinal stromal tumors. Report of the GIST Consensus Conference of 20-21 March 2004, under the auspices of ESMO. Ann Oncol. 2005 Apr;16(4):566-78. doi: 10.1093/annonc/mdi127. PMID 15781488
- [Background] Casali PG, Jost L, Reichardt P, Schlemmer M, Blay JY; ESMO Guidelines Working Group. Gastrointestinal stromal tumors: ESMO clinical recommendations for diagnosis, treatment and follow-up. Ann Oncol. 2008 May;19 Suppl 2:ii35-8. doi: 10.1093/annonc/mdn080. No abstract available. PMID 18456761
- [Background] Demetri GD, Benjamin RS, Blanke CD, Blay JY, Casali P, Choi H, Corless CL, Debiec-Rychter M, DeMatteo RP, Ettinger DS, Fisher GA, Fletcher CD, Gronchi A, Hohenberger P, Hughes M, Joensuu H, Judson I, Le Cesne A, Maki RG, Morse M, Pappo AS, Pisters PW, Raut CP, Reichardt P, Tyler DS, Van den Abbeele AD, von Mehren M, Wayne JD, Zalcberg J; NCCN Task Force. NCCN Task Force report: management of patients with gastrointestinal stromal tumor (GIST)--update of the NCCN clinical practice guidelines. J Natl Compr Canc Netw. 2007 Jul;5 Suppl 2:S1-29; quiz S30. PMID 17624289
- [Background] Reichardt P, Blay JY, Mehren Mv. Towards global consensus in the treatment of gastrointestinal stromal tumor. Expert Rev Anticancer Ther. 2010 Feb;10(2):221-32. doi: 10.1586/era.09.171. PMID 20131998
- [Background] Montemurro M, Schoffski P, Reichardt P, Gelderblom H, Schutte J, Hartmann JT, von Moos R, Seddon B, Joensuu H, Wendtner CM, Weber E, Grunwald V, Roth A, Leyvraz S. Nilotinib in the treatment of advanced gastrointestinal stromal tumours resistant to both imatinib and sunitinib. Eur J Cancer. 2009 Sep;45(13):2293-7. doi: 10.1016/j.ejca.2009.04.030. Epub 2009 May 19. PMID 19467857
- [Background] Sleijfer S, Ray-Coquard I, Papai Z, Le Cesne A, Scurr M, Schoffski P, Collin F, Pandite L, Marreaud S, De Brauwer A, van Glabbeke M, Verweij J, Blay JY. Pazopanib, a multikinase angiogenesis inhibitor, in patients with relapsed or refractory advanced soft tissue sarcoma: a phase II study from the European organisation for research and treatment of cancer-soft tissue and bone sarcoma group (EORTC study 62043). J Clin Oncol. 2009 Jul 1;27(19):3126-32. doi: 10.1200/JCO.2008.21.3223. Epub 2009 May 18. PMID 19451427
- [Background] Freedman LS. Tables of the number of patients required in clinical trials using the logrank test. Stat Med. 1982 Apr-Jun;1(2):121-9. doi: 10.1002/sim.4780010204. PMID 7187087
- [Background] Corless CL, Fletcher JA, Heinrich MC. Biology of gastrointestinal stromal tumors. J Clin Oncol. 2004 Sep 15;22(18):3813-25. doi: 10.1200/JCO.2004.05.140. PMID 15365079
- [Background] Mazur MT, Clark HB. Gastric stromal tumors. Reappraisal of histogenesis. Am J Surg Pathol. 1983 Sep;7(6):507-19. doi: 10.1097/00000478-198309000-00001. PMID 6625048
- [Background] Schaldenbrand JD, Appelman HD. Solitary solid stromal gastrointestinal tumors in von Recklinghausen's disease with minimal smooth muscle differentiation. Hum Pathol. 1984 Mar;15(3):229-32. doi: 10.1016/s0046-8177(84)80184-7. PMID 6421716
- [Background] Nilsson B, Bumming P, Meis-Kindblom JM, Oden A, Dortok A, Gustavsson B, Sablinska K, Kindblom LG. Gastrointestinal stromal tumors: the incidence, prevalence, clinical course, and prognostication in the preimatinib mesylate era--a population-based study in western Sweden. Cancer. 2005 Feb 15;103(4):821-9. doi: 10.1002/cncr.20862. PMID 15648083
- [Background] DeMatteo RP, Lewis JJ, Leung D, Mudan SS, Woodruff JM, Brennan MF. Two hundred gastrointestinal stromal tumors: recurrence patterns and prognostic factors for survival. Ann Surg. 2000 Jan;231(1):51-8. doi: 10.1097/00000658-200001000-00008. PMID 10636102
- [Background] Emile JF. [GIST: definition, physiopathology]. J Chir (Paris). 2008;145 Suppl 3:6S1-3. French. PMID 19060840
- [Background] Hirota S, Ohashi A, Nishida T, Isozaki K, Kinoshita K, Shinomura Y, Kitamura Y. Gain-of-function mutations of platelet-derived growth factor receptor alpha gene in gastrointestinal stromal tumors. Gastroenterology. 2003 Sep;125(3):660-7. doi: 10.1016/s0016-5085(03)01046-1. PMID 12949711
- [Background] Rubin BP, Singer S, Tsao C, Duensing A, Lux ML, Ruiz R, Hibbard MK, Chen CJ, Xiao S, Tuveson DA, Demetri GD, Fletcher CD, Fletcher JA. KIT activation is a ubiquitous feature of gastrointestinal stromal tumors. Cancer Res. 2001 Nov 15;61(22):8118-21. PMID 11719439
- [Background] Heinrich MC, Corless CL, Duensing A, McGreevey L, Chen CJ, Joseph N, Singer S, Griffith DJ, Haley A, Town A, Demetri GD, Fletcher CD, Fletcher JA. PDGFRA activating mutations in gastrointestinal stromal tumors. Science. 2003 Jan 31;299(5607):708-10. doi: 10.1126/science.1079666. Epub 2003 Jan 9. PMID 12522257
- [Background] Fletcher CD, Berman JJ, Corless C, Gorstein F, Lasota J, Longley BJ, Miettinen M, O'Leary TJ, Remotti H, Rubin BP, Shmookler B, Sobin LH, Weiss SW. Diagnosis of gastrointestinal stromal tumors: A consensus approach. Hum Pathol. 2002 May;33(5):459-65. doi: 10.1053/hupa.2002.123545. PMID 12094370
- [Background] Blay JY, Le Cesne A, Ray-Coquard I, Bui B, Duffaud F, Delbaldo C, Adenis A, Viens P, Rios M, Bompas E, Cupissol D, Guillemet C, Kerbrat P, Fayette J, Chabaud S, Berthaud P, Perol D. Prospective multicentric randomized phase III study of imatinib in patients with advanced gastrointestinal stromal tumors comparing interruption versus continuation of treatment beyond 1 year: the French Sarcoma Group. J Clin Oncol. 2007 Mar 20;25(9):1107-13. doi: 10.1200/JCO.2006.09.0183. PMID 17369574
- [Background] Verweij J, Casali PG, Zalcberg J, LeCesne A, Reichardt P, Blay JY, Issels R, van Oosterom A, Hogendoorn PC, Van Glabbeke M, Bertulli R, Judson I. Progression-free survival in gastrointestinal stromal tumours with high-dose imatinib: randomised trial. Lancet. 2004 Sep 25-Oct 1;364(9440):1127-34. doi: 10.1016/S0140-6736(04)17098-0. PMID 15451219
- [Background] Blanke CD, Rankin C, Demetri GD, Ryan CW, von Mehren M, Benjamin RS, Raymond AK, Bramwell VH, Baker LH, Maki RG, Tanaka M, Hecht JR, Heinrich MC, Fletcher CD, Crowley JJ, Borden EC. Phase III randomized, intergroup trial assessing imatinib mesylate at two dose levels in patients with unresectable or metastatic gastrointestinal stromal tumors expressing the kit receptor tyrosine kinase: S0033. J Clin Oncol. 2008 Feb 1;26(4):626-32. doi: 10.1200/JCO.2007.13.4452. PMID 18235122
- [Background] Blanke CD, Demetri GD, von Mehren M, Heinrich MC, Eisenberg B, Fletcher JA, Corless CL, Fletcher CD, Roberts PJ, Heinz D, Wehre E, Nikolova Z, Joensuu H. Long-term results from a randomized phase II trial of standard- versus higher-dose imatinib mesylate for patients with unresectable or metastatic gastrointestinal stromal tumors expressing KIT. J Clin Oncol. 2008 Feb 1;26(4):620-5. doi: 10.1200/JCO.2007.13.4403. PMID 18235121
- [Background] Heinrich MC, Maki RG, Corless CL, Antonescu CR, Harlow A, Griffith D, Town A, McKinley A, Ou WB, Fletcher JA, Fletcher CD, Huang X, Cohen DP, Baum CM, Demetri GD. Primary and secondary kinase genotypes correlate with the biological and clinical activity of sunitinib in imatinib-resistant gastrointestinal stromal tumor. J Clin Oncol. 2008 Nov 20;26(33):5352-9. doi: 10.1200/JCO.2007.15.7461. Epub 2008 Oct 27. PMID 18955458
- [Background] Kumar R, Knick VB, Rudolph SK, Johnson JH, Crosby RM, Crouthamel MC, Hopper TM, Miller CG, Harrington LE, Onori JA, Mullin RJ, Gilmer TM, Truesdale AT, Epperly AH, Boloor A, Stafford JA, Luttrell DK, Cheung M. Pharmacokinetic-pharmacodynamic correlation from mouse to human with pazopanib, a multikinase angiogenesis inhibitor with potent antitumor and antiangiogenic activity. Mol Cancer Ther. 2007 Jul;6(7):2012-21. doi: 10.1158/1535-7163.MCT-07-0193. PMID 17620431
- [Background] Sternberg CN, Davis ID, Mardiak J, Szczylik C, Lee E, Wagstaff J, Barrios CH, Salman P, Gladkov OA, Kavina A, Zarba JJ, Chen M, McCann L, Pandite L, Roychowdhury DF, Hawkins RE. Pazopanib in locally advanced or metastatic renal cell carcinoma: results of a randomized phase III trial. J Clin Oncol. 2010 Feb 20;28(6):1061-8. doi: 10.1200/JCO.2009.23.9764. Epub 2010 Jan 25. PMID 20100962
- [Background] Hutson TE, Davis ID, Machiels JP, De Souza PL, Rottey S, Hong BF, Epstein RJ, Baker KL, McCann L, Crofts T, Pandite L, Figlin RA. Efficacy and safety of pazopanib in patients with metastatic renal cell carcinoma. J Clin Oncol. 2010 Jan 20;28(3):475-80. doi: 10.1200/JCO.2008.21.6994. Epub 2009 Dec 14. PMID 20008644
- [Derived] Mir O, Cropet C, Toulmonde M, Cesne AL, Molimard M, Bompas E, Cassier P, Ray-Coquard I, Rios M, Adenis A, Italiano A, Bouche O, Chauzit E, Duffaud F, Bertucci F, Isambert N, Gautier J, Blay JY, Perol D; PAZOGIST study group of the French Sarcoma Groupe-Groupe d'Etude des Tumeurs Osseuses (GSF-GETO). Pazopanib plus best supportive care versus best supportive care alone in advanced gastrointestinal stromal tumours resistant to imatinib and sunitinib (PAZOGIST): a randomised, multicentre, open-label phase 2 trial. Lancet Oncol. 2016 May;17(5):632-41. doi: 10.1016/S1470-2045(16)00075-9. Epub 2016 Apr 5. PMID 27068858